CLINICAL TRIAL: NCT02790203
Title: Perioperative Use of a Selective COX2 Inhibitor in Patients Undergoing Elective Colorectal Surgery: the Effect on Post-operative Bowel Motility and Post-operative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Nir Horesh resident Department of Surgery and Transplant, Resident in General Surgery, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2913-16-SMC
Record Dates: First submitted 2016-05-22; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Prevention of Post Operative Ileus
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib (Experimental): Celecoxib will be given orally to patients participating in the study and allocated to the treatment group, for an intervention period of 6 days, starting from the day of surgery.
  Celecoxib will be given throughout the intervention period of the study orally at a dose of 400 mg per day divided into two doses, a dose which is within the recommended and a widely used dosage and is expected to induce a significant inhibition of prostaglandin synthesis by the COX2 pathway. Celecoxib will be given throughout the intervention period of the study orally at a dose of 400 mg per day divided into two doses.
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Placebo will be given orally to patients participating in the study and allocated to the control group that will receive placebo, for an intervention period of 6 days, starting from the day of surgery.
  Placebo will be given throughout the intervention period of the study orally in capsules that resemble the drug, twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — NSAIDS
  Arms: Celecoxib
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Perioperative Celecoxib to promote bowel movement and to reduce post-operative pain after elective colonic resection.

DETAILED DESCRIPTION:
Post-operative ileus is a common surgical complication occurring in with up to 20% of patients, with a significant clinical and economical effect.

Many preventative measures have been tested to promote gastrointestinal motility following intestinal surgery have been suggested.

The medical intervention in the proposed study includes administration of a selective COX-2 inhibitor, specifically Celecoxib, in the peri-operative period following an elective colon resection. Celecoxib is a nonsteroidal anti-inflammatory drug (NSAID) with anti-inflammatory, analgesic, and antipyretic therapeutic effects.

The drug is approved for use in by the ministry of health in Israel and in the United states. The study aims to assess the use of this widely used medication for evaluation of the clinical effect on post-operative bowel transit, as well as the drugs' effect on post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18 and 80
* Patients planned for elective colorectal surgery with primary anastomosis
* ASA score of 1-3
* Patients that are able to sign an informed consent and comply with the protocol

Exclusion Criteria:

* Patients with inflammatory bowel disease
* Patients that require emergency surgery
* Patients with renal failure, measured by Creatinine level > 1.5 mg/dL (>106.1 micro mol/l)
* Patients with significant liver failure (known cirrhosis, Bilirubin level>2 mg/dL or 34.2 µmol/L)
* Patients with known allergy to any medication from the non-steroidal anti-inflammatory drug group.
* Patients treated chronically with any type of COX inhibitor.
* Patients treated with NSAIDS including Aspirin 7 days prior to the date of surgery.
* Patients with active peptic disease
* Patient expected to take muscle relaxants, tricyclic antidepressants, tranquilizers, sedatives, hypnotics or neuroleptics in the postoperative period
* Patient with dysphagia or that have a difficulty swallowing capsules or tablets, or is unable to tolerate oral medication
* Pregnant / lactating women.
* Patients participating in any other interventional clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
First flatus/bowel movement (questionnaire) | 48 to 72 hours after surgery
  Reduction of time for first flatus/bowel movement from 48 hours to 72 hours in average following surgery.

SECONDARY OUTCOMES:
Reduction of post operative ileus (questionnaire) | First week after surgery
  Reduction of post-operative ileus rate in patients following colorectal surgery, treated with Celecoxib when compared with patients treated with placebo.
Post operative pain reduction (VAS score) | First week after surgery
  Post-operative pain reduction quality in patients treated with Celecoxib when compared with patients treated with placebo following surgery.
Reduction of opoids consumption (registration of all medications) | First month after surgery
  Reduction the amount of opioids consumed in patients treated with Celecoxib when compared with patients treated with placebo following surgery.
Post operative complication rate (patients follow up) | First month after surgery
  Post-operative complication rate, more specifically the rate of anastomotic leakage in patients treated with Celecoxib compared with patients treated with placebo.

IPD SHARING:
Plan to Share IPD: Undecided